CLINICAL TRIAL: NCT00354536
Title: A Single-blinded Randomized, Placebo-controlled, Staggered-parallel, Escalating-dose Study to Investigate the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of Subcutaneous Injections of GSK 716155 in Subjects With Type 2 Diabetes Mellitus
Brief Title: In-patient Study With GSK716155 In Patients With Type 2 Diabetes Mellitus
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: GLP106073
Record Dates: First submitted 2006-07-18; First posted 2006-07-20 (Estimated); Last update posted 2016-10-26 (Estimated); Status verified 2016-10

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: GSK716155; albiglutide; pharmacodynamics; pharmacokinetics
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Who Masked: Participant

ARMS (2):
- albiglutide (Active Comparator): albiglutide injection
  Interventions: Drug: GSK716155 subcutaneous injections
- albiglutide placebo (Placebo Comparator): placebo injection
  Interventions: Biological: placebo injection

INTERVENTIONS:
Drug: GSK716155 subcutaneous injections — albiglutide subcutaneous injection
  Arms: albiglutide
Biological: placebo injection — placebo injection
  Other Names: placebo
  Arms: albiglutide placebo

SUMMARY:
This study is a placebo-controlled study in patients with Type 2 Diabetes Mellitus to assess safety and tolerability parameters, the levels of GSK716155 in the bloodstream when it is given at the same dose 7 days apart, and the impact this medication has on various substances in the blood. Assessments include ECGs, vital signs, repeat blood sampling and monitoring of any side effects.

ELIGIBILITY:
Inclusion criteria:

* Subjects must have type 2 diabetes mellitus that has been diagnosed for at least three months.
* Must be taking either (1) no medication for their diabetes or (2) taking metformin, a sulfonylurea, or metformin and a sulfonylurea.
* Subjects must be willing to wash-out of these medications for 14 days prior to the start of the study.
* Subjects must have a BMII between 25 and 40 kg/m² and weigh at leas 50kg.
* Women must be of non-childbearing potential.

Exclusion criteria:

* Laboratory values that meet certain criteria (for example, total cholesterol > 240 mg/dL).
* Clinically significant hepatic enzyme elevation.
* Fasting plasma glucose greater than 240mg/dL.
* Positive test result for Hepatitis B surface antigen, positive Hepatitis C or HIV.
* Any major illness other than diabetes.
* Previous use of insulin as treatment for diabetes.
* Significant renal disease as defined by screening lab tests.
* History of drug or other allergy, which in the opinion of the investigator contradicts subject participation.
* Smoking or use of nicotine-containing products within the previous 6 months.
* History of alcohol or drug abuse.
* Unwilling to abstain from alcohol during the study.
* Unwilling to abstain from caffeine- or xanthine-containing products during the study.
* Use of St. John's Wort during the study.
* Has donated 500 nL or more blood within 56 days of dosing or plans to donate blood in the month following study participation.
* Previously received any GLP-1 mimetic that has moe than 70% sequence homology to GLP-1.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2006-02; Primary Completion 2006-09 (Actual); Study Completion 2006-09 (Actual)

PRIMARY OUTCOMES:
blood plasma levels of GSK716155 | on days 2 & 9

SECONDARY OUTCOMES:
blood plasma levels of GSK716155 | on days 2 & 9

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (5):
- United States (5):
  - GSK Investigational Site, Miramar, Florida
  - GSK Investigational Site, Orlando, Florida
  - GSK Investigational Site, Honolulu, Hawaii
  - GSK Investigational Site, Portland, Oregon
  - GSK Investigational Site, San Antonio, Texas

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Derived] Young MA, Wald JA, Matthews JE, Scott R, Hodge RJ, Zhi H, Reinhardt RR. Clinical pharmacology of albiglutide, a GLP-1 receptor agonist. Postgrad Med. 2014 Nov;126(7):84-97. doi: 10.3810/pgm.2014.11.2836. PMID 25387217
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Clinical Study Report: GLP106073 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: GLP106073 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: GLP106073 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: GLP106073 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: GLP106073 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: GLP106073 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: GLP106073 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register